CLINICAL TRIAL: NCT07050680
Title: Assessment of Bioaccessibility of Oat Bioactive Compounds and Contaminants in Human Volunteers
Brief Title: How Healthy Are Your Oats?
Acronym: HISU_101
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2-037-25
Record Dates: First submitted 2025-06-19; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Mycotoxin Biomonitoring
Keywords: Human exposure; Toxicokinetics; Urinary excretion
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oat intervention arm (Experimental): All participants will consume a single dose of an oat test meal
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Single dose of commercially available Oat food test meal

SUMMARY:
Oat foods are commonly consumed as healthy breakfast options and their nutritional value is well recognised. Oats are a rich source of fibre, micronutrients and non-nutrient bioactive compounds, but at the same time cereals including oats can be contaminated with mycotoxins. To fully understand the nutritional benefits and potential food safety risks of oat consumption, this study aims to assess the nutritional composition of an oat food and the bioavailability of bioactive oat constituents and their metabolite profile in urine of volunteers consuming a single portion of an oat breakfast. This study requires 16 healthy volunteers to consume one portion of oats and collect their urine over 48 hours after the test meal. No other sample collection is required.

DETAILED DESCRIPTION:
Cereal foods are important part of a healthy, balanced diet. Amongst cereals, oats form an important part of a Scottish diet and are an important agricultural commodity. Oats are well-known for their high nutritional value containing high-quality fatty acids (oleic and linoleic acids), proteins with high amino acid profiles and dietary fibre, most namely in the form of soluble β-glucans. These β-glucans have well-documented health benefits regarding cholesterol-lowering effects in humans. In addition to macronutrients, oats are also a rich source of micronutrients including tocopherols and a range of minerals. As such, the consumption of oats is highly recommended by dietary advice. However, oats and other cereals are also known to be at risk of contamination with naturally occurring fungal toxins called mycotoxins. Previous studies have demonstrated the presence of detectable levels of mycotoxins formed by Fusarium fungi in oat crops and oat foods. Current risk assessments by the European Food Safety Authority and the UK Food Standard Agency aim to establish maximum permitted levels of these mycotoxins in foods. The maximum levels aim to protect consumers from high level exposure and potential health effects.

Rationale for Study This study is part of a wider programme of work investigating the health benefits and potential food safety risks of oats. The presence of phytochemicals and Fusarium mycotoxins in oat foods has been confirmed and the bioaccessibility of these bioactive compounds in the human gut has been demonstrated in-vitro. To fully quantify dietary exposure of individuals to these bioactive compounds, detailed work is needed to understand the rate of bioaccessibility of bioactive compounds from oat foods and their absorption and excretion into urine in humans. This detailed information will inform future studies aimed at assessing dietary exposure and risk.

The proposed study aims to feed a single dose of an oat food to healthy volunteers. The study will assess how the oat food is digested and the bioactive compounds absorbed and excreted in vivo. The food will be selected to contain low and safe mycotoxin levels.

ELIGIBILITY:
Inclusion Criteria:

Adult males and females (aged 18 - 65 years) who are healthy with a BMI in the normal to overweight range (18.5-29.9)

Exclusion Criteria:

* Anyone who currently suffers from gastrointestinal or metabolic diseases, liver disease or kidney disease
* Anyone who currently has an eating disorder (anorexia, bulimia, binge eating, night eating syndrome)
* Anyone who is taking prescribed medication related to gastrointestinal, metabolic, liver or kidney disease
* Anyone who has taken antibiotics in the past 3 months
* Anyone who is allergic or intolerant to oat foods
* Anyone who is currently pregnant or breastfeeding
* Anyone who is currently taking vitamin or mineral supplements (unless they agree to discontinue supplementation 2 weeks before the study)
* Anyone currently participating in another research study
* Anyone who is unable to fluently speak, read and understand English
* Anyone who is unable to give written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Kinetics of mycotoxin absorption and excretion | Hourly urine sample collection up to 16 hours post-intervention, then bulk urine collection at 24 and 48 hours.
  Urinary excretion profile of oat-derived mycotoxins and metabolites will be assessed after consumption of a single oat-based test meal in 16 volunteers. Volunteers will collect hourly urine samples. Samples will be analysed for mycotoxin metabolites using established LC-MS/MS methodology.

CONTACTS AND LOCATIONS:
Locations (1):
- Rowett Institute, University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No